CLINICAL TRIAL: NCT00568386
Title: Acute Comfort and Blurring Profile Evaluation Comparing Systane Lubricant Eye Drops to Optive Lubricant Eye Drops
Brief Title: Acute Comfort and Blur of Systane and Optive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M-07-02
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Results first posted 2010-03-10 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: Dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Systane Lubricant Eye Drops (Experimental): Systane Lubricant Eye Drops 1 drop in each eye one time
  Interventions: Other: Systane Lubricant Eye Drops
- Optive Lubricant Eye Drops (Active Comparator): Optive Lubricant Eye Drops 1 drop each one time
  Interventions: Other: Optive Lubricant Eye Drops

INTERVENTIONS:
Other: Systane Lubricant Eye Drops — Systane Lubricant Eye Drops 1 drop each eye once time
  Arms: Systane Lubricant Eye Drops
Other: Optive Lubricant Eye Drops — Optive Lubricant Eye Drops 1 drop each eye one time
  Arms: Optive Lubricant Eye Drops

SUMMARY:
To evaluate drop comfort, acceptability, preference and blur profile between two marketed artificial tears in both dry eye and non-dry eye patient population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, normal eyes OR documented diagnosis of dry eye

Exclusion Criteria:

* Must not have worn contact lenses for 7 days preceding enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-11; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Christensen, Principal Investigator — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical Clinic Nov. 2007
Pre-assignment Details: 24 hr. wash out between treatment periods
Groups:
- Systane Drops Then Optive Drops: Systane Drops then Optive Drops
- Optive Drops Then Systane Drops: Optive Drops then Systane Drops
Period: Overall Study
Arm/Group | Systane Drops Then Optive Drops | Optive Drops Then Systane Drops
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Systane Drops Then Optive Drops | Optive Drops Then Systane Drops | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Visual Blur
Description: Visual blur profile is a visual scale ranging from 0 (no blur) to 50 (most blurry). Patients were asked to rate there vision on a specific focal point (an object in the room) through 3 minutes.
Time Frame: 3 minutes post dose
Measure: Mean (Full Range); unit: Units on a scale
Groups:
- Systane Lubricant Eye Drops: Systane lubricant eye drops
- Optive Lubricant Eye Drops: Optive Lubricant eye drops
Arm/Group | Systane Lubricant Eye Drops | Optive Lubricant Eye Drops
Number analyzed (Participants) | 40 | 40
Units on a scale | 27.7 [0 to 49] | 33.55 [10 to 50]

ADVERSE EVENTS:
Arm/Group | Systane Lubricant Eye Drops | Optive Lubricant Eye Drops
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No